CLINICAL TRIAL: NCT01455519
Title: True Functional Restoration and Analgesia in Non-Radicular Low Back Pain: a Prospective Double Blind, Placebo-controlled Study of Hydromorphone ER
Brief Title: True Functional Restoration and Analgesia in Non-Radicular Low Back Pain
Acronym: Covidien
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shirley Ryan AbilityLab (Other)
Collaborators: Mallinckrodt (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RIC_Cov_2011
Record Dates: First submitted 2011-10-11; First posted 2011-10-20 (Estimated); Results first posted 2015-07-13 (Estimated); Last update posted 2017-10-24 (Actual); Status verified 2017-10

CONDITIONS: Low Back Pain
Keywords: Low Back Pain; Back Pain; Chronic back pain
MeSH Terms: conditions — Low Back Pain; Back Pain | interventions — Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sugar pill (Placebo Comparator): Subjects may receive a pill with no medicine.
  Interventions: Drug: Sugar pill
- Hydromorphone ER (Active Comparator): Subjects received study drug: Hydromorphone ER
  Interventions: Drug: Hydromorphone ER

INTERVENTIONS:
Drug: Hydromorphone ER — Total target dose of 32 mg/day. All subjects will have a lead in for 2 weeks; then begin a 'forced' 2-week up-titration schedule as follows: 8mg/d (1 pill, 5 days), 16mg mg/d (2 pills, 5 days), and 24mg/d (3 pills, 5 days) then finally 32 mg/d (4 pills a day) for the 'stable dose' phase of the study, or identical placebo pills. If intolerable side effects occur, the dose may be reduced to last tolerable does, a minimum of 8 mg/day (or one pill a day), at the discretion of the PI. Subjects unable to tolerate 8 mg/day will be discontinued from the study. A 2-week down-titration will be used.
  Other Names: Exalgo(hydromorphone HCl), CII (77605306)
  Arms: Hydromorphone ER
Drug: Sugar pill — Sugar pill
  Arms: Sugar pill

SUMMARY:
You are asked to take part in this study because you have chronic, non-radicular low back pain. This study is done to investigate the pain relieving effects of the study drug Exalgo (Hydromorphone ER) for people who experience chronic non-radicular low back pain. The purpose of this research is to look at how the study drug can be used to benefit people who experience this type of pain. This is a phase IV study done to study the safety and effectiveness of the drug. At this point the drug has been approved by the Food and Drug Administration and has been studied in more than 2,000 pain patients in clinical trials, including individuals with low back pain. About 36 subjects will take part in this study.

DETAILED DESCRIPTION:
As a participant in this study, you will be asked to come to the Rehabilitation Institute of Chicago (RIC), Center for Pain Studies (446 E Ontario St. Suite 1011, Chicago, IL 60611). Your part in this study will last for 8 weeks and will involve 3 visits to the Rehabilitation Institute of Chicago and anywhere from weekly phone calls to phone calls every other day.

If you are in this study, you will be placed in one of two study groups: one group will receive the study drug and one will receive a placebo. You will be assigned a study group by chance using a process similar to the flip of a coin. This process is called randomization. Neither you nor the study staff will select the group you will be in. A placebo looks like the study drug but is an inactive substance that has no medication. Researchers use a placebo to see if the study drug works better or is safer than not taking anything. You will have a 66% chance of getting the study drug. You will receive placebo at some point during the study but you will not know whether you are receiving placebo or study drug during the entire study. However, if you have a medical emergency, the investigators can get this information.

ELIGIBILITY:
Inclusion Criteria:

* Meets our criteria for Chronic Non-Radicular Back Pain (CNRBP): non-radiating (below buttocks), no frank weakness or atrophy, no sensory or reflex changes
* If female, is not pregnant or breast feeding, and not currently attempting to conceive; if of childbearing potential, use of a highly effective method of birth control (as determined by Pl).
* Able to read and speak English and provide informed consent; ages: 18-90.
* Able to understand and comply with all data collection methodology.
* Subjects may continue any non opioid, non acetaminophen stable drug regimen with no changes during the course of study and not use rescue medications 12 hours before testing.
* Subjects taking opioids must agree to detoxify for the protocol. If they agree they will detox under the direction of the PI before entering the protocol. They may begin the acetaminophen rescue med as per the protocol while in detox.
* Must have pain greater than or equal to 5 on a 10 point Numeric Rating scale (NRS) at phone screening, or pain greater than or equal to 50 on VAS at visit one.

Exclusion Criteria:

* Subjects with hypersensitivity to Opioids, Acetominophen or Exalgo.
* Subjects with severe or untreated psychiatric disturbance (e.g. mania, depression [esp suicidality], anxiety, substance dependence).
* Subjects with a clinical diagnosis of fibromyalgia or polymyalgia rheumatica.
* Subjects with severe ongoing or unaddressed medical conditions (e.g. Renal or Hepatic disease [creatinine>1.5 ml/dl; AST or ALT> 3x normal limit], uncontrolled hypertension), pulmonary disease, uncontrolled seizure disorder, gastoparesis or urinary retention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2011-10; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Norman Harden, M.D., Principal Investigator — Shirley Ryan AbilityLab
Locations (1):
- Rehabilitation Institute of Chicago, Chicago, Illinois, United States

REFERENCES:
- See also: Site Contact Information — http://www.ric.org/research/centers/pain/index.aspx

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 51 subjects were enrolled at baseline. 13 withdrew from the study after visit 1, and 3 no longer met criteria at visit 2.
Groups:
- Hydromorphone ER: Hydromorphone ER Hydromorphone ER: Total target dose of 32 mg/day. All subjects will have a lead in for 2 weeks; then begin a 'forced' 2-week up-titration schedule as follows: 8mg/d (1 pill, 5 days), 16mg mg/d (2 pills, 5 days), and 24mg/d (3 pills, 5 days) then finally 32 mg/d (4 pills a day) for the 'stable dose' phase of the study, or identical placebo pills. If intolerable side effects occur, the dose may be reduced to last tolerable does, a minimum of 8 mg/day (or one pill a day), at the discretion of the PI. Subjects unable to tolerate 8 mg/day will be discontinued from the study. A 2-week down-titration will be used.
Period: Overall Study
Arm/Group | Sugar Pill | Hydromorphone ER
Started | 12 | 23
Completed | 8 | 18
Not Completed | 4 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sugar Pill | Hydromorphone ER | Total
Number analyzed (Participants) | 12 | 23 | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.8 (10.7) | 46.6 (9.2) | 47.7 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 12 | 17
  Male | 7 | 11 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 10 | 23 | 33
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 13 | 21
  White | 1 | 8 | 9
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 2 | 2 | 4
Body Mass Index [Mean (Standard Deviation); unit: kg/m2] | 32.8 (10.4) | 29.3 (8.4) | 30.5 (9.1)
Duration of Pain [Mean (Standard Deviation); unit: years] | 12.6 (12.3) | 8.7 (7.8) | 10.0 (9.3)

OUTCOME MEASURES:

1. Primary Outcome: Change in McGill Pain Questionnaire - Short Form
Description: The McGill Pain Questionnaire - Short Form (MPQ-SF) is a well-validated pain measure that permits separation of the sensory and affective components of pain, which are added together to compute a total score. The scale ranges from 0-45 (0=no pain, 45=the most pain).
Time Frame: Collected at 2 visits over 8-10 weeks: Visit 1 and Visit 4. Change values were calculated from Baseline to post intervention
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Sugar Pill | Hydromorphone ER
Number analyzed (Participants) | 8 | 18
units on a scale | -0.73 (2.33) | -3.78 (1.7)

2. Primary Outcome: Change in VAS
Description: Visual Analogue Scale is a self report pain scale on a scale 0(no pain) to 100 (the worst pain imaginable).
Time Frame: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Sugar Pill | Hydromorphone ER
Number analyzed (Participants) | 8 | 18
units on a scale | -10.57 (9.54) | -10.67 (6.91)

3. Secondary Outcome: Change in PASS
Description: Anxiety scores were collected at least two data points. The Pain Anxiety Symptoms Scale (PASS) is a scale from 0 - 100, where 0 = no anxiety and 100 = the most anxiety.
Time Frame: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Sugar Pill | Hydromorphone ER
Number analyzed (Participants) | 8 | 18
units on a scale | -7.14 (2.94) | -5.85 (2.21)

4. Secondary Outcome: Change in Pain Disability
Description: The Pain Disability Index (PDI) is a seven-item, validated instrument that assesses perceived disability in seven key life areas. It provides a total disability score, and is an indirect measure of self efficacy. The Pain Disability Scale is a scale from 0 - 70, where 0 = no Disability and 70 = the most Disability.
Time Frame: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Sugar Pill | Hydromorphone ER
Number analyzed (Participants) | 8 | 18
units on a scale | -9.84 (4.56) | -9.25 (3.36)

5. Secondary Outcome: Change in Stair Climb Time
Description: Time to climb 1 flight of stairs
Time Frame: as for outcome 1
Measure: Mean (Standard Error); unit: seconds
Arm/Group | Sugar Pill | Hydromorphone ER
Number analyzed (Participants) | 8 | 18
seconds | 1.28 (1.08) | -1.25 (0.8)

6. Secondary Outcome: Change in Treadmill Distance Walked
Description: Treadmill distance walked in 6 minutes
Time Frame: as for outcome 1
Measure: Mean (Standard Error); unit: miles
Arm/Group | Sugar Pill | Hydromorphone ER
Number analyzed (Participants) | 8 | 18
miles | 0.02 (0.02) | 0.02 (0.01)

7. Secondary Outcome: Change in Sit to Stand Repetitions
Description: Sit to stand repetitions completed in 1 minute
Time Frame: as for outcome 1
Measure: Mean (Standard Error); unit: number of repetitions
Arm/Group | Sugar Pill | Hydromorphone ER
Number analyzed (Participants) | 8 | 18
number of repetitions | -1.07 (1.52) | .54 (1.14)

8. Secondary Outcome: Change in Distance to Floor
Description: Distance from fingers to Floor when bending forward. A functional test of flexibility
Time Frame: as for outcome 1
Measure: Mean (Standard Error); unit: centimeters
Arm/Group | Sugar Pill | Hydromorphone ER
Number analyzed (Participants) | 8 | 18
centimeters | -4.61 (3.03) | -4.02 (2.26)

9. Secondary Outcome: Change in Time to Lift Box
Description: Time to lift 13 pound box to floor and back up to table.
Time Frame: as for outcome 1
Measure: Mean (Standard Error); unit: seconds per lift
Arm/Group | Sugar Pill | Hydromorphone ER
Number analyzed (Participants) | 8 | 18
seconds per lift | -1.45 (1.13) | -1.06 (0.8)

10. Secondary Outcome: Change in NRS After Stair Climb
Description: Numeric Rating Scale (NRS) pain score was given verbally after completing functional stair climb test on a scale 0-10 (0=none, and 10=the worst).
Time Frame: as for outcome 1
Measure: Mean (Standard Error); unit: NRS pain score
Arm/Group | Sugar Pill | Hydromorphone ER
Number analyzed (Participants) | 8 | 18
NRS pain score | 0.04 (0.23) | -0.11 (0.17)

11. Secondary Outcome: Change in NRS After Treadmill Walk
Description: Numeric Rating Scale (NRS) pain score was given verbally after completing functional treadmill walk test on a scale 0-10 (0=none, and 10=the worst).
Time Frame: as for outcome 1
Measure: Mean (Standard Error); unit: NRS pain score
Arm/Group | Sugar Pill | Hydromorphone ER
Number analyzed (Participants) | 8 | 18
NRS pain score | 0.1 (0.44) | -0.51 (0.32)

12. Secondary Outcome: Change in NRS After Sit to Stand Repetitions
Description: Numeric Rating Scale (NRS) pain score was given verbally after completing functional sit to stand test on a scale 0-10 (0=none, and 10=the worst).
Time Frame: as for outcome 1
Measure: Mean (Standard Error); unit: NRS pain score
Arm/Group | Sugar Pill | Hydromorphone ER
Number analyzed (Participants) | 8 | 18
NRS pain score | -0.24 (0.34) | -0.57 (0.25)

13. Secondary Outcome: Change in NRS After Box Lift
Description: Numeric Rating Scale (NRS) pain score was given verbally after completing functional box lift test on a scale 0-10 (0=none, and 10=the worst).
Time Frame: as for outcome 1
Measure: Mean (Standard Error); unit: NRS pain score
Arm/Group | Sugar Pill | Hydromorphone ER
Number analyzed (Participants) | 8 | 18
NRS pain score | 0.39 (0.58) | -0.43 (0.36)

ADVERSE EVENTS:
Arm/Group | Sugar Pill | Hydromorphone ER
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/23
Other Adverse Events (participants affected / at risk) | 5/12 | 15/23
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sugar Pill (N=12) | Hydromorphone ER (N=23)
nausea (General disorders) | 0 | 6
fatigue (General disorders) | 0 | 4
drowsiness (General disorders) | 1 | 9
vomiting (General disorders) | 1 | 2
trouble sleeping (General disorders) | 0 | 1
itchiness (General disorders) | 2 | 1
dizziness (General disorders) | 0 | 1
stomach pain (Gastrointestinal disorders) | 1 | 0
diarrhea (General disorders) | 0 | 1
ear infection (Ear and labyrinth disorders) | 0 | 1
lack of appetite (General disorders) | 0 | 1
heartburn (Gastrointestinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No